CLINICAL TRIAL: NCT06564571
Title: Artificial Intelligence in Endoscopic Ultrasound
Status: Recruiting | Type: Observational
Sponsor: Orlando Health, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 24.015.01
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2024-08

CONDITIONS: Pancreatic Cancer; Pancreas Disease; Pancreatic Cyst
Keywords: pancreatic disease; pancreatic cancer; pancreatic cyst; artificial intelligence
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Diseases; Pancreatic Cyst

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients undergoing endoscopic ultrasound procedures: Patients will undergo endoscopic ultrasound procedures as planned. Abnormalities in the pancreas identified by the endoscopist during the endoscopic ultrasound examination will be correlated against those detected by the AI platform.
  Interventions: Device: Patients undergoing endoscopic ultrasound procedures

INTERVENTIONS:
Device: Patients undergoing endoscopic ultrasound procedures — Patients will undergo endoscopic ultrasound procedures as planned. Abnormalities in the pancreas identified by the endoscopist during the endoscopic ultrasound examination will be correlated against those detected by the AI platform.

SUMMARY:
The objective of the study is to determine if this artificial intelligence system is capable of detecting abnormalities in the pancreas that are identified by an endoscopist at endoscopic ultrasound procedures.

DETAILED DESCRIPTION:
Endoscopic Ultrasound (EUS) is an equipment where an ultrasound transducer is attached to the tip of the endoscope. When advanced to the stomach the organs outside such as the pancreas and liver can be visualized in great detail. This enables diagnosis of conditions such as pancreatic cancer. However, an endoscopist must undergo training to accurately interpret these ultrasound images.

The investigators are in the process of developing an artificial intelligence system that could potentially interpret EUS images. The objective of the study is to determine if this artificial intelligence system is capable of detecting abnormalities in the pancreas that are identified by an endoscopist at endoscopic ultrasound procedures. Such correlation if established will lead to possible development of an artificial intelligence platform that can diagnose pancreatic diseases. Such development will potentially minimize human error and decrease learning curve to gain proficiency in EUS.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Any patient undergoing endoscopic ultrasound examination

Exclusion Criteria:

* Age < 18 years

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient 18 years or over undergoing endoscopic ultrasound examination
Sampling Method: Non-Probability Sample
Enrollment: 310 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Rate of detection pancreatic abnormalities by AI | 1 day
  Ability of AI to detect pancreatic abnormalities as identified by an endoscopist during EUS examination of the pancreas.

SECONDARY OUTCOMES:
Rate of detection pancreatic solid mass lesions by AI | 1 day
  Ability of AI to detect pancreatic solid mass lesions as identified by an endoscopist during EUS examination of the pancreas.
Rate of detection pancreatic cystic lesions by AI | 1 day
  Ability of AI to detect pancreatic cystic lesions as identified by an endoscopist during EUS examination of the pancreas.

CONTACTS AND LOCATIONS:
Overall Officials: Shyam Varadarajulu, MD, Principal Investigator — Orlando Health, Digestive Health Institute
Locations (1):
- Orlando Health, Orlando, Florida, United States